CLINICAL TRIAL: NCT01038115
Title: A Randomised Study Comparing Pulmonary Vein Isolation Using the Occluding Cryoballoon, Conventional Radiofrequency Energy, or Both in the Treatment of Atrial Fibrillation (AF).
Brief Title: Study Comparing Pulmonary Vein Isolation With the Cryoballoon, Radiofrequency Energy, or Both in the Treatment of Atrial Fibrillation (AF)
Acronym: Cryo Vs RFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005841
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2011-03

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (3):
- Cryoballoon (Active Comparator)
  Interventions: Procedure: Atrial fibrillation ablation
- Radiofrequency (Active Comparator)
  Interventions: Procedure: Atrial fibrillation ablation
- Cryoballoon + Radiofrequency together (Active Comparator)
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Comparison of three different techniques for pulmonary vein isolation

SUMMARY:
The purpose of this study is to perform a prospective, randomised study investigating the safety and efficacy of cryoballoon catheter ablation compared with radiofrequency ablation, or both together in the treatment of paroxysmal AF.

The hypotheses for this study are (1) that cryothermal energy is as effective and safe as using radiofrequency energy in the treatment of paroxysmal AF and is associated with a better long term outcome, and (2) that use of both cryothermy and RF in combination is as effective and safe as using either radiofrequency energy or cryothermy alone and is associated with a better long term outcome.

DETAILED DESCRIPTION:
Pulmonary vein isolation is an important treatment for patients with atrial fibrillation (AF), particularly those in whom antiarrhythmic drugs are ineffective or cannot be tolerated. One method involves the use of radiofrequency energy and 3-D mapping system to produce a series of lesions (small burn areas) within the heart. Another method involves passing a balloon (called a cryoballoon) into the heart and freezing the parts of the heart muscle that the veins drain into. Both methods appear to be effective from known data. However, it is not known if use of either method alone or both together is the most effective. We aim to perform a prospective, randomized clinical trial comparing these three strategies.

Substudy 1: Use of cardiac MRI to evaluate ablation lesions. Some patients will also be asked to undergo an MRI scan of the heart before the ablation procedure, and again at three months and one year following the procedure. This will allow us to examine the potential role for MRI in imaging scar tissue formed by the ablation, and help us understand the time course of scar formation and changes to that part of the heart following the ablation.

Substudy 2: Platelet reactivity and activation in AF, and the impact of curative ablation. Blood and urine samples will be taken pre- and 3 months post ablation to see if platelet reactivity and activation are affected by AF compared to established normal ranges, and whether curative ablation impacts on this.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented paroxysmal AF on at least 2 occasions and accepted for catheter ablation.

Exclusion Criteria

* Significant valvular disease
* Previous left atrial ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2008-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Freedom from AF after a single procedure at 12 months. | 12 months
  Freedom from AF or any other atrial tachyarrhythmia lasting > 30 seconds (symptomatic or not) at 12 months following a single ablation procedure.

SECONDARY OUTCOMES:
Complication rates, costs, fluoroscopy times, radiation exposure, and long term success. MRI substudy: sensitivity & specificity for determining ablation lesions. Platelet substudy: Platelet activation post ablation compared to baseline. | 0-12 months post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and the London NHS Trust, London, London, United Kingdom

REFERENCES:
- [Derived] Hunter RJ, Baker V, Finlay MC, Duncan ER, Lovell MJ, Tayebjee MH, Ullah W, Siddiqui MS, McLEAN A, Richmond L, Kirkby C, Ginks MR, Dhinoja M, Sporton S, Earley MJ, Schilling RJ. Point-by-Point Radiofrequency Ablation Versus the Cryoballoon or a Novel Combined Approach: A Randomized Trial Comparing 3 Methods of Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation (The Cryo Versus RF Trial). J Cardiovasc Electrophysiol. 2015 Dec;26(12):1307-14. doi: 10.1111/jce.12846. Epub 2015 Nov 25. PMID 26727045